CLINICAL TRIAL: NCT00501254
Title: Randomised Clinical Trial, Parallel, Double Blind, to Evaluate the Influence of the ASA-SR (Slow-Release) in the Platelet Parameters and the Oxidative Status, in Patients With Coronary Disease of Chronic Evolution During 12 Months
Brief Title: Pharmacodynamic Trial, of Slow Release ASA, in Platelet Functionalism, a Long Term Treatment Period
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Rottapharm Spain (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TROM-EC-ECC-01; EudraCT number: 2004-000398-76
Record Dates: First submitted 2007-07-13; First posted 2007-07-16 (Estimated); Last update posted 2007-07-18 (Estimated); Status verified 2007-07

CONDITIONS: Cardiovascular Disease
Keywords: Slow release ASA; Platelet functionalism; Secondary cardiovascular prevention
MeSH Terms: conditions — Cardiovascular Diseases

INTERVENTIONS:
Drug: Slow release acetyl salicylic acid
Behavioral: Antithrombotic effect

SUMMARY:
Evaluation of the pharmacodynamic profile (antiaggregant profile, balance of prostanoids and nitric oxid) of a ASA-SR (slow-release)formulation in comparison with a ASA NR (normal release), 150 mg, during 12 months of treatment.

DETAILED DESCRIPTION:
* A large clinical trials have established the efficacy of the antiaggregant products in patients with ischemic cardiopathy, stroke and intermittent claudication.
* The acetylsalicylic acid (ASA) is the most used antiaggregant substance, nevertheless, and spite of being centenarian, it last some questions pending regarding the most appropriate dose, mechanisms of action implicated, the association with oder drugs, and the pharmaceutical fom in order to improve the efficacy and safety of the ASA.
* Some previous studies indicate that the slow release form of ASA has a different behaviour in the platelet effect in comparison with plain formulation.
* The aim of this study is to demonstrate the best antiaggregant and safety profile of a low dose of a slow release formulation in a long term treatment period of one year.

ELIGIBILITY:
Inclusion Criteria:

* Previous episodes of myocardial infarction
* Previous episodes of instable angina pectoris
* Previous coronary revascularization
* Significant arterial coronary disease

Exclusion Criteria:

* Patients with other pathologies that require treatment with other antiaggregants
* Patients in treatment with low molecular weight heparin or oral anticoagulants
* Patients with antecedents of hypersensibility to ASA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-02; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The evaluation of the effect of treatment with slow release ASA on the tromboxane/prostacyclin balance and its repercusion in the platelet aggregation | one year

SECONDARY OUTCOMES:
Safety profile of the two different formulations of ASA (Slow Release and Normal Release) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Eloy Rueda, MD, Principal Investigator — Hosp. Universitario Virgen de la Victoria, Málaga (Spain); José Pedro de la Cruz, MD, phD, Principal Investigator — Departamento de Farmacología y Terapéutica Clínica Facultad de Medicina, Universidad de Málaga; José Antonio González Correa, MD, phD, Principal Investigator — Departamento de Farmacología y Terapéutica Clínica Facultad de Medicina, Universidad de Málaga
Locations (1):
- Hospital Universitario Virgen de la Victoria, Málaga, Málaga, Spain